CLINICAL TRIAL: NCT00096083
Title: A Phase II Study Of Hepatic Arterial Infusion Of Melphalan With Venous Filtration Via Peripheral Hepatic Perfusion (PHP) For Unresectable Primary And Metastatic Cancers Of The Liver
Brief Title: Hepatic Arterial Infusion of Melphalan With Hepatic Perfusion in Treating Patients With Unresectable Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Delcath Systems Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000391827; NCI-04-C-0273; NCI-6332; DELCATH-G990039; NCT00091455 (obsolete NCT alias)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Cancer
Keywords: advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; liver metastases; adenocarcinoma of the colon; adenocarcinoma of the esophagus; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the gallbladder; adenocarcinoma of the pancreas; adenocarcinoma of the rectum; adenocarcinoma of the stomach; carcinoma of the appendix; recurrent gallbladder cancer; unresectable gallbladder cancer; recurrent colon cancer; stage IV colon cancer; recurrent esophageal cancer; stage IV esophageal cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent gastric cancer; stage IV gastric cancer; recurrent rectal cancer; stage IV rectal cancer; small intestine adenocarcinoma; recurrent small intestine cancer; recurrent islet cell carcinoma; recurrent pheochromocytoma; metastatic pheochromocytoma; pulmonary carcinoid tumor; thyroid gland medullary carcinoma; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; recurrent pancreatic cancer; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; stage IV pancreatic cancer; intraocular melanoma; conjunctival melanoma; iris melanoma; recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Colonic Neoplasms; Adenocarcinoma Of Esophagus; Rectal Neoplasms; Appendiceal Neoplasms; Gallbladder Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Stomach Neoplasms; Carcinoma, Islet Cell; Pheochromocytoma; Carcinoma, Medullary; Pancreatic Neoplasms; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma; Uveal Melanoma; Melanoma | interventions — Melphalan

ARMS (1):
- Melphalan Administration PHP (Active Comparator)
  Interventions: Drug: isolated perfusion; Drug: melphalan

INTERVENTIONS:
Drug: isolated perfusion
Drug: melphalan

SUMMARY:
RATIONALE: Hepatic arterial infusion uses a catheter to deliver anticancer substances directly into the liver. Drugs used in chemotherapy, such as melphalan, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving an hepatic arterial infusion of melphalan together with hepatic perfusion works in treating patients with unresectable liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate and duration of response in patients with unresectable primary or metastatic liver cancer treated with intrahepatic arterial infusion of melphalan with venous filtration via peripheral hepatic perfusion.

Secondary

* Determine the patterns of recurrence in patients treated with this regimen.
* Determine progression-free and overall survival of patients treated with this regimen.
* Evaluate the safety and tolerability of this regimen in these patients.
* Assess the filter characteristics including melphalan pharmacokinetics and filtration of cytokines and clotting factors during and after treatment.

OUTLINE: Patients are stratified according to primary tumor histology (neuroendocrine tumor vs primary hepatic malignancy vs adenocarcinoma of gastrointestinal or other origin).

Patients undergo peripheral isolated hepatic perfusion in which a catheter is placed via the groin into the hepatic artery and another into the hepatic vein. Patients then receive melphalan as an intrahepatic arterial infusion over 15-30 minutes. Treatment repeats approximately every 3-8 weeks for up to 6 total infusions in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 105 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatic malignancy

  * Unresectable disease
  * Disease predominantly in the parenchyma of the liver
  * One of the following primary tumor histologies:

    * Adenocarcinoma of gastrointestinal or other origin
    * Neuroendocrine tumor (except gastrinoma)
    * Primary hepatic malignancy (e.g., hepatocellular cancer or intra-hepatic cholangiocarcinoma)
    * Cutaneous or ocular melanoma (patients must have received prior regional melphalan therapy)
  * Hepatic metastases from colorectal tumors allowed provided patient has undergone prior first-line chemotherapy, including irinotecan or oxaliplatin
* Limited unresectable extrahepatic disease on preoperative radiological studies allowed if life-limiting component of progressive disease is in the liver

  * Limited extrahepatic disease includes, but is not limited to, the following:

    * Up to 4 pulmonary nodules each < 1 cm in diameter
    * Retroperitoneal lymph nodes each < 3 cm in diameter
    * Less than 10 skin or subcutaneous metastases each < 1 cm in diameter
    * Asymptomatic bone metastases that have been or could be palliatively treated with external beam radiotherapy
    * Resectable solitary metastasis to any site
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 16 and over

Sex

* Male or Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 75,000/mm^3
* Hematocrit > 27%
* Absolute neutrophil count ≥ 1,300/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* PT ≤ 2 seconds of upper limit of normal (ULN)
* AST and ALT ≤ 10 times ULN
* No Childs class B or C cirrhosis
* No portal hypertension by history, endoscopy, or radiologic studies

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No congestive heart failure
* LVEF ≥ 40%

Pulmonary

* No chronic obstructive pulmonary disease
* FEV_1 ≥ 30% of predicted
* DLCO ≥ 40% of predicted

Immunologic

* No active infection
* No severe allergic reaction to iodine contrast agent that is not controlled by premedication with antihistamines or steroids
* No known hypersensitivity reaction to melphalan or heparin in the presence of a heparin induced thrombocytopenia (HIT) antibody

Other

* Weight > 35 kg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No documented latex allergy
* No evidence of intracranial abnormalities which would lead to risk for bleeding with anticoagulation (e.g., stroke or active metastasis)
* No evidence of active ulcer disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 month since prior biologic therapy and recovered

Chemotherapy

* See Disease Characteristics
* More than 1 month since prior chemotherapy and recovered

Endocrine therapy

* Premenopausal women (i.e., have had a period within the past 12 months) must be willing to undergo hormonal suppression during study treatment

Radiotherapy

* See Disease Characteristics
* More than 1 month since prior radiotherapy and recovered

Surgery

* No prior Whipple resection

Other

* Prior intrahepatic perfusion (with or without arterial infusion with floxuridine) or peripheral hepatic perfusion allowed provided the patient had a radiographic partial response of 3 months' duration after therapy
* No concurrent immunosuppressive drugs
* No concurrent chronic anticoagulation therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the response rate and duration of response to intra-hepatic infusion of melphalan with subsequent venous hemofiltration in patients with primary and metastatic hepatic malignancies | Survivial

SECONDARY OUTCOMES:
To determine the patterns of recurrence following percutaneous hepatic perfusions (PHP) with melphalan | Survival
To determine the progression free and overall survival in patients with hepatic malignancies following this therapy | Survivial

CONTACTS AND LOCATIONS:
Overall Officials: Marybeth Hughes, MD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States